CLINICAL TRIAL: NCT05533476
Title: Multi Sensory Stimulation And Priming (MuSSAP) in Infants (4-12 Months of Age) at Risk of Developing Unilateral Cerebral Palsy (uCP)
Brief Title: Multi Sensory Stimulation And Priming (MuSSAP) in Infants at Risk of Unilateral Cerebral Palsy
Acronym: MuSSAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sint Maartenskliniek (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 724; NL52823.091.15 (Other: CCMO)
Record Dates: First submitted 2022-09-05; First posted 2022-09-09 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Unilateral Cerebral Palsy
Keywords: Cerebral Palsy; Multisensory Stimulation; Hand function; Infants; Early intervention
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multi Sensory Stimulation And Priming (Experimental): 8 weeks, 30 minutes per day home based MuSSAP training.
  Interventions: Behavioral: Multi Sensory Stimulation and Priming
- Intensive Usual Care (Upper Limb) (Experimental): 8 weeks, 30 minutes per day home based Intensive Usual Care (Upper Limb).
  Interventions: Behavioral: Intensive Usual Care (Upper Limb)

INTERVENTIONS:
Behavioral: Multi Sensory Stimulation and Priming — In the MuSSAP intervention group, the infant wears a multisensory stimulating wristband aiming at increasing attention for the affected upper limb and readiness to initiate a goal-directed movement. Parents are instructed to present a toy to their child if the child shows attention to the affected arm and hand. Upper extremity motor activities like reaching, grasping and holding are practiced. Parents practice daily and once a week the training will be guided or conducted by a physical or occupational therapist in the home environment. An occupational therapist from the rehabilitation center will coach parents during the intervention period through the internet, by means of analyzing the videos from the home training.
  Arms: Multi Sensory Stimulation And Priming
Behavioral: Intensive Usual Care (Upper Limb) — The Intensive Usual Care (Upper Limb) intervention is a more intensive (in duration and frequency) version of standard Usual Care with focus on the motor development of the affected upper extremity. Upper extremity motor activities like reaching, grasping and holding are practiced. Parents practice daily and once a week the training will be guided or conducted by a physical or occupational therapist in the home environment. An occupational therapist from the rehabilitation center will coach parents during the intervention period through the internet, by means of analyzing the videos from the home training.
  Arms: Intensive Usual Care (Upper Limb)

SUMMARY:
A pilot randomized clinical trial exploring the effect of a Multi Sensory Stimulation And Priming (MuSSAP) training on improving manual ability in infants at risk of developing unilateral Cerebral Palsy.

DETAILED DESCRIPTION:
Rationale:

Unilateral Cerebral Palsy (uCP) results from early brain damage. In adults, brain damage in one side of the (pre) motor cortex is associated with functional problems in the contralateral side of the body and vice versa. This is related to extensive crossings of the descending corticospinal tracts connecting the central motor systems with the musculature of the extremities. However, during the first years of our lives, crossings of the corticospinal tracts are less defined and the motor system relies on both ipsi- and contralateral connections to control the extremities. In children with uCP the classical development and strengthening of the crossed connections of the corticospinal tracts might be hampered. Although reorganization with ipsilateral corticospinal tracts can mediate useful hand function, patients with the most favourable functional outcome retain crossed projections from the affected hemisphere. To facilitate maturation of the corticospinal tracts, it seems crucial to start early with intervention at the stage that the corticospinal tracts show high plasticity. Attention benefits from multisensory congruent signals, particularly if this congruency involves rhythmical similarity. Attention influences the sensitivity of neurons to detect sensory activity and the ability of neurons to detect sensory stimulation. Formation of neural pathways is facilitated by increasing activity in (new) functional neural circuits. During the multisensory stimulation, motor actions of both or one arm and hand will be provoked. In contrast to the functional training focused primarily on motor output, MuSSAP enhances motor learning by stimulating the perception-action loop. In this study, we propose to pilot test whether a new intervention; Multi Sensory Stimulation And Priming (MuSSAP) can be applied in clinical practice in infants 4-12 months of age with diagnosed unilateral cerebral damage having increased risk on the development of unilateral cerebral palsy.

Objective:

Primary objective: The following hypothesis will be tested: MuSSAP in infants 4-12 months of age with diagnosed unilateral cerebral damage, is a feasible protocol and results in an enhanced motor development as compared to Intensive Usual Care (Upper Limb).

Secondary Objective(s): Assessment of feasibility of the intervention: Can the MuSSAP intervention and procedures be successfully executed and delivered to the participants? Assessment of acceptability: Suitability of the intervention and the study procedures from the perspective of the participants. Determining effect sizes for a future full-scale randomized clinical trial and clinical relevance.

Study design:

The study is designed as a pilot randomized clinical trial (RCT) with three measuring moments (before intervention, after intervention, and follow-up).

Study population:

The study population consists of 16 infants at risk for developing unilateral cerebral palsy. These infants will either be born preterm suffering from unilateral periventricular haemorrhagic infarction, or born at term suffering from unilateral middle cerebral artery (MCA) stroke. The infants at risk will be allocated either to the MuSSAP intervention group (8 infants) or the Intensive Usual Care (Upper Limb) group (8 infants) by randomisation. Data of 8 typically developing infants will be used to monitor typical development of infants of 4-12 months old.

Intervention:

Both the MuSSAP and the Intensive Usual Care (Upper Limb) interventions are home based and consist of 30 minutes (divided in 3 periods of 10 minutes each) of remediating impairments practicing specific age related movements and skills, each day for an 8-week period, conducted by the parents and once a week by a physical or occupational therapist in the home environment. Upper extremity motor activities like reaching, grasping and holding are practiced. Coaching of parents and therapists will be performed by the occupational therapist of the Sint Maartenskliniek. This will be realised through analysing video recordings of the intervention in the home environment once a week.

Multi Sensory Stimulation And Priming (MuSSAP): In the MuSSAP intervention a custom made wristband will be used to provide rhythmical congruent multisensory stimulations to the affected arm and hand aiming to increase attention for the affected upper limb. Subsequently, motor actions of the affected arm and hand will be provoked.

Intensive Usual Care (Upper Limb): This intervention is a more intensive (in duration and frequency) version of standard Usual Care with focus on the motor development of the affected upper extremity.

In both intervention groups infants will additionally receive pediatric physical therapy in the home environment (usual care) focusing on gross motor development.

Primary study parameters/outcome of the study:

The primary study parameter aims at development of handfunction/ manual ability (measured with the Hand Assessment for Infants (HAI)).

ELIGIBILITY:
Inclusion Criteria Intervention:

* Born preterm suffering from unilateral periventricular haemorrhagic infarction with involvement of the corticospinal tracts
* Born term suffering from unilateral middle cerebral artery stroke with involvement of the corticospinal tracts
* ±4 months of age (time the infant starts to reach with at least one hand) to 10 months of age (age corrected in case of prematurity)

Exclusion Criteria Intervention:

* Severe epilepsy
* Severe sensory impairments (blindness, deafness)
* Children with clinical signs of bilateral involvement
* Inability of parents to respond to interviews or questionnaires in Dutch
* Expected inability of parents to adhere to the home-based protocol

Inclusion Criteria age matched typical developing infants:

* Born term (≥37 weeks gestational age)
* Birth weight within a normal range (≥2500 grams)

Exclusion Criteria age matched typical developing infants:

* Inability of parents to respond to interviews or questionnaires in Dutch
* Expected inability of parents to adhere to planned measuring moments

Ages: 4 Months to 10 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2016-06-14 (Actual); Primary Completion 2018-08-20 (Actual); Study Completion 2018-08-20 (Actual)

PRIMARY OUTCOMES:
Mean change from T0 in manual ability as assessed by the Hand Assessment for Infants (HAI) | T0 (before the start of the intervention), T1 (after the 8-week intervention), T2 (8 weeks after the interventions stops)
  The HAI is intended to evaluate the quality of goal-directed manual actions in infants, 3-12 months of age, at risk of developing unilateral CP. The test procedure comprises a semi-structured video-recorded 10-15-min play session. HAI is intended to detect and quantify possible asymmetry between hands by providing scores for each hand separately (Each Hand sum Score (EaHS) (range 0-24)), and to provide a measure of bilateral hand use (Both Hands Measure (BoHM) (range 0-100)) with a higher score reflecting a better outcome.
Adherence based on total training time | During 8 week intervention
  Parents fill out a digital time registration form to assess intervention adherence every day. Adherence will be calculated by dividing the registrated total training time by total planned training time (28 hours).

SECONDARY OUTCOMES:
Motor development as assessed by the Bayley Scales of Infant and Toddler Development - Third Edition (Dutch version) (Bayley-III-NL) | T0 (before the start of the intervention), T1 (after the 8-week intervention), T2 (8 weeks after the interventions stops)
  The motor scale of the Bayley-III-NL will be used to assess motor development. The gross motor (GM) subscale raw scores (range 0-72) will be determined on all assessment points, the fine motor (FM) subscale raw scores (range 0-66) on T0 only. A higher score reflects a better outcome.
Gross motor development as assessed by the Gross Motor Function Measure (GMFM) | T0 (before the start of the intervention), T1 (after the 8-week intervention), T2 (8 weeks after the interventions stops)
  The GMFM contains eighty-eight items grouped into five dimensions (e.g. lying and rolling, sitting, crawling and kneeling, standing, walking, running and jumping) and is sensitive to motor developmental changes over time.
Quality of life as assessed by the Infant and Toddler Quality of life Questionnaire (ITQOL) | T0 (before the start of the intervention), T1 (after the 8-week intervention), T2 (8 weeks after the interventions stops)
  The infant/toddler quality of life questionnaire (ITQOL) is a generic parent-completed 'profile-measure' for health status and health-related quality of life of children between 2 months and 5 years old. Raw scale scores are transformed to a standardized 0-100 continuum with a higher score reflecting a better health status.
Reaction time of self-initiated goal-directed movement and attention as assessed by the Video Observation Attention Affected Hand (VOAAH) | During 8 week intervention
  The VOAAH is a video-observation tool that is used to assess time to self-initiated goal-directed movement and time to attention. Training session videos recorded by parents are manually scored using a standardized protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Pauline Aarts, PhD, Principal Investigator — Sint Maartenskliniek

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Verhaegh AP, Nuijen NB, Aarts PB, Nijhuis-van der Sanden MWG, Willemsen MA, Groen BE, Vriezekolk JE. Parents' experiences with a home-based upper limb training program using a video coaching approach for infants and toddlers with unilateral cerebral palsy: a qualitative interview study. BMC Pediatr. 2022 Jun 29;22(1):380. doi: 10.1186/s12887-022-03432-w. PMID 35768858
- [Derived] Verhaegh APM, Groen BE, Aarts PBM, van Ee R, Willemsen MAAP, Jongsma MLA, Nijhuis-van der Sanden MWG. Multisensory Stimulation and Priming (MuSSAP) in 4-10 Months Old Infants with a Unilateral Brain Lesion: A Pilot Randomised Clinical Trial. Occup Ther Int. 2023 Jan 6;2023:8128407. doi: 10.1155/2023/8128407. eCollection 2023. PMID 36711188
- See also: Medical Ethical Registration and Reviewing form — https://www.toetsingonline.nl/to/ccmo_search.nsf/fABRpop?readform&unids=2005C3E3527D170FC1258611001B9157
- See also: Website information infant and toddler upper limb rehabilitation programs Sint Maartenskliniek — https://www.maartenskliniek.nl/kinderzorg/kinderrevalidatie/arm-en-handrevalidatie-voor-baby-s-en-peuters